CLINICAL TRIAL: NCT00759746
Title: Childhood Obesity Treatment: A Maintenance Approach
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Seattle Children's Hospital (Other); University of Florida (Other); State University of New York at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201107083; 2R01HD036904 (NIH)
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Childhood Overweight; Childhood Obesity
Keywords: Weight loss maintenance
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weight Maintenance Education (Active Comparator): Participants assigned to this group will receive the Weight Maintenance Education intervention. They will meet every other week during the maintenance phase of the study for a total of 16 sessions over 8 months. During the visit, participants will participate in a series of interactive workshops within child and parent groups to learn general information about healthy eating and physical activity.
  Interventions: Behavioral: Weight Maintenance Education
- SFM+ Low Dose (Experimental): Participants assigned to this group will receive the SFM+ Low Dose.
  Interventions: Behavioral: SFM+ Low Dose
- SFM+ High Dose (Experimental): Participants assigned to this group will receive the SFM+ High Dose.
  Interventions: Behavioral: SFM+ High Dose

INTERVENTIONS:
Behavioral: SFM+ Low Dose — The SFM intervention assumes people need a social environment that supports changes in eating and physical activity for continued weight maintenance. Therefore, the SFM intervention will focus on helping families create a social environment that supports weight maintenance (e.g., children being friends with physically active peers). Participants in this group will meet less often than families that receive the Social Facilitation Maintenance (SFM) - High Dose intervention, giving them more opportunities to practice new skills between clinic visits.
  Arms: SFM+ Low Dose
Behavioral: Weight Maintenance Education — The Weight Maintenance Education intervention will help participants in parent and child groups to learn more about healthy eating and physical activity in a group setting. Participants will also learn about exercise and exercise safety, hydration during exercise, and stress management. Parent and child groups will combine for particular on-site and off-site activities, such as cooking demonstrations, grocery store tours, gym tours, and dance lessons.
  Arms: Weight Maintenance Education
Behavioral: SFM+ High Dose — The SFM intervention assumes people need a social environment that supports changes in eating and physical activity for continued weight maintenance. Therefore, the SFM intervention will focus on helping families create a social environment that supports weight maintenance (e.g., children being friends with physically active peers). Participants in this group will meet more often than families that receive the Social Facilitation Maintenance (SFM) - Low Dose intervention, allowing for more in-depth discussion and practice of key skills and concepts related to creating a social environment that supports a healthy lifestyle. These participants will receive more feedback and reinforcement from fellow group members, family interventionists, and group leaders for practicing their new behaviors.
  Arms: SFM+ High Dose

SUMMARY:
The purpose of this study is to determine the effect of dose and content of an enhanced weight maintenance treatment on children's ability to maintain weight loss following a standard weight loss treatment.

DETAILED DESCRIPTION:
Childhood Obesity (CO) prevalence in the United States has tripled in recent decades, and nearly 30% of children aged 6 to 11 are overweight or obese. CO is a serious public health problem, and is associated with both immediate and long-term health problems (e.g., hypertension, type 2 diabetes, asthma) and psychosocial problems (e.g., social isolation, depression, eating disorder symptomatology). Furthermore, CO is a significant risk factor for adult obesity with several prospective studies showing that, if untreated, about half of overweight grade-school children remain obese as adults. Fortunately, children respond favorably to family-based behavioral weight loss treatment (FBT), the most well-established intervention for the treatment of overweight in children 7 to 12 years old. Weight loss treatments for overweight children have been associated with significant physical and psychosocial health benefits; however, despite initial success with lifestyle interventions, considerable relapse often occurs once treatment ends. Clearly, CO is a significant public health problem, and long-term maintenance of weight loss remains a priority to stem the increased costs to the individual and society. Therefore, we propose to conduct a multi-site randomized controlled trial with overweight children (N=241) and their parents (N=241) [for a total N=482]. All participants will complete 4 months of FBT and then be randomized to one of three, 8-month maintenance conditions: (1) Weight Maintenance Therapy, who will receive SFM - Low Dose [LOW] (16 sessions over 8 months), (2) Intensive Weight Maintenance Therapy, who will receive SFM - High Dose [HIGH] (32 sessions over 8 months), or (3) Current Standard of Care, who will receive Weight Maintenance Education (16 sessions over 8 months). Relative weight and associated outcomes will be assessed at 0 (pre-weight loss), 4 (post-weight loss), 12 (post-maintenance treatment),18 months and 24 months. Additionally, brief assessments will be conducted at four points during the course of maintenance treatment to measure presumed mediators.

ELIGIBILITY:
Inclusion Criteria:

* Children will be between the ages of 7 and 11 and at or above the 85th percentile for weight.
* At least one parent of the participating child must be overweight (BMI ≥ 25).
* One parent must agree to attend all parent/child treatment meetings as the participating parent.
* Participants must be able to speak and comprehend English.

Exclusion Criteria:

* Participating parent or child having a thought disorder, suicidality, bipolar disorder, or drug or alcohol dependence.
* Participating parent or child having a physical disability or illness that prevents performance of physical activity at level equivalent to a brisk walk or that places severe restriction on diet.
* Participating parent or child being on a medication regimen that affects weight.
* Participating parent or child being involved in active psychiatric treatment for an ongoing problem that causes either social or occupational impairment.
* Parents (participating and nonparticipating) and children having an eating disorder (i.e., anorexia nervosa, bulimia nervosa, binge eating disorder) or having subclinical levels of eating disturbance (i.e., reporting key eating disorder behaviors of purging, fasting, or binge eating more than two times per month).

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 482 (Actual)
Dates: Start 2009-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Child percent overweight | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Denise E Wilfley, PhD, Principal Investigator — Washington University School of Medicine; Brian Saelens, Ph.D., Principal Investigator — Seattle Children's Hospital
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Seattle Children's Hospital Research Institute, Seattle, Washington

REFERENCES:
- [Result] Hayes JF, Altman M, Kolko RP, Balantekin KN, Holland JC, Stein RI, Saelens BE, Welch RR, Perri MG, Schechtman KB, Epstein LH, Wilfley DE. Decreasing food fussiness in children with obesity leads to greater weight loss in family-based treatment. Obesity (Silver Spring). 2016 Oct;24(10):2158-63. doi: 10.1002/oby.21622. Epub 2016 Sep 7. PMID 27601189
- [Result] Altman M, Cahill Holland J, Lundeen D, Kolko RP, Stein RI, Saelens BE, Welch RR, Perri MG, Schechtman KB, Epstein LH, Wilfley DE. Reduction in food away from home is associated with improved child relative weight and body composition outcomes and this relation is mediated by changes in diet quality. J Acad Nutr Diet. 2015 Sep;115(9):1400-7. doi: 10.1016/j.jand.2015.03.009. Epub 2015 May 8. PMID 25963602
- [Result] Holland JC, Kolko RP, Stein RI, Welch RR, Perri MG, Schechtman KB, Saelens BE, Epstein LH, Wilfley DE. Modifications in parent feeding practices and child diet during family-based behavioral treatment improve child zBMI. Obesity (Silver Spring). 2014 May;22(5):E119-26. doi: 10.1002/oby.20708. Epub 2014 Mar 25. PMID 24458836
- [Result] Best JR, Theim KR, Gredysa DM, Stein RI, Welch RR, Saelens BE, Perri MG, Schechtman KB, Epstein LH, Wilfley DE. Behavioral economic predictors of overweight children's weight loss. J Consult Clin Psychol. 2012 Dec;80(6):1086-1096. doi: 10.1037/a0029827. Epub 2012 Aug 27. PMID 22924332
- [Derived] Fowler LA, Litt MD, Rotman SA, Conlon RPK, Jakubiak J, Stein RI, Balantekin KN, Welch RR, Perri MG, Epstein LH, Wilfley DE. Relation of social network support to child health behaviors among children in treatment for overweight/obesity. Eat Weight Disord. 2022 Jun;27(5):1669-1678. doi: 10.1007/s40519-021-01303-4. Epub 2021 Sep 21. PMID 34549372
- [Derived] Grammer AC, Best JR, Fowler LA, Balantekin KN, Stein RI, Conlon RPK, Saelens BE, Welch RR, Perri MG, Epstein LH, Wilfley DE. General and Eating Disorder Psychopathology in Relation to Short- and Long-Term Weight Change in Treatment-Seeking Children: A Latent Profile Analysis. Ann Behav Med. 2021 Jun 28;55(7):698-704. doi: 10.1093/abm/kaaa076. PMID 32914852
- [Derived] Fowler LA, Grammer AC, Ray MK, Balantekin KN, Stein RI, Kolko Conlon RP, Welch RR, Perri MG, Epstein LH, Wilfley DE. Examining the interdependence of parent-child dyads: Effects on weight loss and maintenance. Pediatr Obes. 2021 Jan;16(1):e12697. doi: 10.1111/ijpo.12697. Epub 2020 Jul 28. PMID 32720457
- [Derived] Rotman SA, Fowler LA, Ray MK, Stein RI, Hayes JF, Kolko RP, Balantekin KN, Engel A, Saelens BE, Welch RR, Perri MG, Epstein LH, Wilfley DE. Family Encouragement of Healthy Eating Predicts Child Dietary Intake and Weight Loss in Family-Based Behavioral Weight-Loss Treatment. Child Obes. 2020 Apr;16(3):218-225. doi: 10.1089/chi.2019.0119. Epub 2019 Dec 12. PMID 31829732
- [Derived] Wilfley DE, Saelens BE, Stein RI, Best JR, Kolko RP, Schechtman KB, Wallendorf M, Welch RR, Perri MG, Epstein LH. Dose, Content, and Mediators of Family-Based Treatment for Childhood Obesity: A Multisite Randomized Clinical Trial. JAMA Pediatr. 2017 Dec 1;171(12):1151-1159. doi: 10.1001/jamapediatrics.2017.2960. PMID 29084318
- [Derived] Balantekin KN, Hayes JF, Sheinbein DH, Kolko RP, Stein RI, Saelens BE, Hurst KT, Welch RR, Perri MG, Schechtman KB, Epstein LH, Wilfley DE. Patterns of Eating Disorder Pathology are Associated with Weight Change in Family-Based Behavioral Obesity Treatment. Obesity (Silver Spring). 2017 Dec;25(12):2115-2122. doi: 10.1002/oby.22028. Epub 2017 Oct 6. PMID 28984076